CLINICAL TRIAL: NCT03818360
Title: Implementation of an Evidence-based Smoking Cessation Intervention Comprising Brief Advice Plus Active Referrals for Smokers Attending Emergency Departments in Hong Kong
Brief Title: Deliver an Evidence-based Smoking Cessation Intervention for Smokers Attending A&E Departments in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 19-032
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Smoking; Smoking Cessation; Evidence-Based Nursing; Emergency Service, Hospital
Keywords: Smoking cessation intervention; Evidence-based; Brief advice; Active referrals; Emergency departments
MeSH Terms: conditions — Smoking; Smoking Cessation; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smokers attending A&E (Experimental): Receive an evidence-based smoking cessation intervention comprising brief advice plus active referrals for smokers attending emergency departments in Hong Kong.
  Interventions: Behavioral: an evidence-based smoking cessation intervention comprising brief advice plus active referrals

INTERVENTIONS:
Behavioral: an evidence-based smoking cessation intervention comprising brief advice plus active referrals — The trained healthcare professionals will be encouraged to deliver brief smoking cessation advice based on the AWARD model to smokers who attend emergency departments and are triaged as semi-urgent or non-urgent. The trained healthcare professionals will ask the smokers their smoking history, then deliver the warning message to the smokers. If the smokers refuse to quit immediately, the trained healthcare professionals will advise them to reduce the number of cigarettes smoked per day, with the goal of complete cessation within 6 months. The healthcare professionals will then actively refer smokers to the chosen service provider within 1 week of recruitment. Smokers will receive proactive telephone calls from the service providers, receive a leaflet about the health-related hazards of smoking and benefits of quitting, and a pocket-sized information card containing brief information about the existing smoking cessation services in Hong Kong.

SUMMARY:
This project aims to deliver an evidence-based smoking cessation intervention comprising the provision of brief cessation advice to smokers attending emergency departments and active referral to existing smoking cessation services. The objectives are as follows:

1. To promote this evidence-based project to emergency departments in various hospitals under the Hospital Authority
2. To construct a network with non-governmental organisations (NGOs) to provide smoking cessation services
3. To train healthcare professionals to use the AWARD model to deliver brief cessation advice to smokers
4. To deliver brief cessation advice via healthcare professionals and actively refer smokers to existing smoking cessation services.

DETAILED DESCRIPTION:
Smoking exerts harmful effects on nearly every organ of the body and is considered responsible for 7 million deaths worldwide every year.1 Despite a decrease in the prevalence of daily cigarette smoking from 23.3% in 1982 to 10.0% in 2017, 615,000 daily smokers2 remain in Hong Kong, where 400,000 hospitalisations per year are attributable to smoking.3 These statistics cannot be overlooked or undervalued.

The provision of medical attention to smokers in physical discomfort who visit accident and emergency departments (AEDs) could be an excellent teachable model, as it provides an invaluable opportunity to encourage smoking cessation. Smokers who consult physicians in an emergency setting are more likely to adopt better health-related behaviours. According to the Hospital Authority,4 approximately 2 million people visit AEDs in Hong Kong each year; of them, 68% are triaged as semi-urgent (level 4) or non-urgent (level 5). The average waiting time for a medical consultation varies among AEDs but generally exceeds 30 min for triage level 4 and 1-2 h for level 5. These wait times represent a golden opportunity in which healthcare professionals could advise smokers to quit and provide information about available smoking cessation programmes.4 However, cigarette smoking is addictive, and cessation is a difficult process associated with a high rate of relapse, particularly among smokers with a high level of nicotine dependency.5 According to the latest Hong Kong Thematic Household Survey, 31.2% of participating cigarette smokers had tried but failed to quit smoking.2 Therefore, an innovative intervention is needed and should be evaluated with the intent to enhance its effectiveness and potential for implementation in clinical settings. Based on the health needs of the community, we propose that such a smoking cessation strategy should combine different components, such as the administration of brief advice by healthcare professionals and the provision of referrals and follow-up boosters by community smoking cessation services, to achieve a larger intervention effect.

Most existing cessation programmes, including stage-matched interventions6 and motivational interviews,7 generally require implementation periods exceeding 30 minutes. Previous reviews have indicated that a comprehensive intervention might more effectively promote smoking cessation, compared to brief advice.8-10 However, the provision of a comprehensive smoking cessation intervention is not feasible in the busy clinical settings of Hong Kong. Indeed, healthcare professionals most commonly cite a lack of time as the reason for their inability to help patients with smoking cessation; specifically, these professionals are very busy and cannot spare even a few extra minutes.11 Other barriers to assistance include a lack of training and experience, lack of confidence in the effectiveness of the interventions and deficiencies in or a lack of incentives, support or requirements from hospital management regarding the implementation of these programmes. Moreover, our previous smoking cessation projects in an outpatient clinical setting revealed that many patients were too impatient to participate in a long intervention, while others expressed a reluctance to participate because of concerns that they might miss or experience delays in their medical consultations or other medical procedures.11-13 Nevertheless, although a brief intervention is more feasible in a clinical setting, it may be too brief and inadequate to have a significant effect on smokers.12,13 Moreover, the effectiveness of some brief interventions for smokers which focus mainly on providing self-help materials is undermined by a failure to offer or arrange any follow-up.9 Evidence indicates that smoking cessation services, including telephone quitlines, are an effective means of supporting smoking cessation efforts.14 However, these services are generally poorly utilised, with a usage rate of 23.2% among smokers in Hong Kong.2 Therefore, the combination of brief cessation advice plus referrals for smokers to utilise existing smoking cessation services in Hong Kong may comprise an alternative strategy that could enhance the effects of intervention, particularly for patients requiring additional counselling.

Interventions will include:

1. Use of brief smoking cessation interventions by healthcare professionals
2. Self-determination intervention for smoking cessation (i.e., immediate or progressive cessation with the ultimate goal of completion over an acceptable period)
3. Active referral

Service targets

Phase I: To promote our project to the emergency departments of hospitals under the Hospital Authority.

Phrase II: To recruit healthcare professionals from participating emergency departments to attend a half-day training workshop.

Phrase III: To provide brief smoking cessation advices by healthcare professionals to smokers who attend emergency departments and actively refer them to existing smoking cessation services

ELIGIBILITY:
* Healthcare professionals employed in the emergency departments of various hospitals under the Hospital Authority
* Smokers attending emergency departments who are triaged as semi-urgent (level 4) or non-urgent (level 5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1603 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Biochemically validated abstinence of smokers at the 6-month follow-up | at the 6-month follow-up
  The self-reported quitters at the 6-month follow-up will be invited to participate in a biochemical validation (measurement of exhaled [CO] and salivary cotinine level). The criteria for validated abstinence are an exhaled CO level of less than 4 ppm and a saliva cotinine level of less than 10 ng/ml.

SECONDARY OUTCOMES:
Biochemically validated abstinence of smokers at the 12-month follow-up | at the 12-month follow-up
  The self-reported quitters at the 12-month follow-up will be invited to participate in a biochemical validation (measurement of exhaled [CO] and salivary cotinine level). The criteria for validated abstinence are an exhaled CO level of less than 4 ppm and a saliva cotinine level of less than 10 ng/ml.
Self-reported 7-day point prevalence of abstinence at the 6-month follow-up | at the 6-month follow-up
  Smokers will be asked to report self-reported 7-day point prevalence of abstinence at the 6-month follow-up
Self-reported 7-day point prevalence of abstinence at the 12-month follow-up | at the 12-month follow-up
  Smokers will be asked to report self-reported 7-day point prevalence of abstinence at the 12-month follow-up
Self-reported reduction of ≥ 50% in cigarette consumption at the 6-month follow-up | at the 6-month follow-up
  Smokers will be asked to report self-reported reduction of ≥ 50% in cigarette consumption at the 6-month follow-up
Self-reported reduction of ≥ 50% in cigarette consumption at the 12-month follow-up | at the 12-month follow-up
  Smokers will be asked to report self-reported reduction of ≥ 50% in cigarette consumption at the 12-month follow-up

OTHER OUTCOMES:
Number of emergency departments participated at the end of recruitment | at 10 months
  Number of emergency departments that agree to join this project
Knowledge of the risk of smoking in trained healthcare professionals before the training workshops | baseline
  The trained healthcare professionals will be asked about their knowledge of the risk of smoking prior to the training workshops
Knowledge of the risk of smoking in trained healthcare professionals at the end of the training workshops | up to 1 week
  The trained healthcare professionals will be asked about their knowledge of the risk of smoking at the end of the training workshops
Knowledge of the risk of smoking in trained healthcare professionals at the 3-month follow-up | at the 3-month follow-up
  The trained healthcare professionals will be asked about their knowledge of the risk of smoking at the 3-month follow-up
Knowledge of the risk of smoking in trained healthcare professionals at the 6-month follow-up | at the 6-month follow-up
  The trained healthcare professionals will be asked about their knowledge of the risk of smoking at the 6-month follow-up
Attitudes towards smoking, tobacco control and smoking cessation in trained healthcare professionals before the training workshops | Baseline
  The trained healthcare professionals will be asked about their attitudes towards smoking, tobacco control and smoking cessation prior to the training workshops
Attitudes towards smoking, tobacco control and smoking cessation in trained healthcare professionals at the end of the training workshops | up to 1 week
  The trained healthcare professionals will be asked about their attitudes towards smoking, tobacco control and smoking cessation at the end of the training workshops
Attitudes towards smoking, tobacco control and smoking cessation in trained healthcare professionals at the 3-month follow-up | at the 3-month follow-up
  The trained healthcare professionals will be asked about their attitudes towards smoking, tobacco control and smoking cessation at the 3-month follow-up
Attitudes towards smoking, tobacco control and smoking cessation in trained healthcare professionals at the 6-month follow-up | at the 6-month follow-up
  The trained healthcare professionals will be asked about their attitudes towards smoking, tobacco control and smoking cessation at the 6-month follow-up
Practices of delivering smoking cessation advice in trained healthcare professionals before the training workshops | baseline
  The trained healthcare professionals will be asked about their practices of delivering smoking cessation advice prior to the training workshops
Practices of delivering smoking cessation advice in trained healthcare professionals at the end of the training workshops | up to 1 week
  The trained healthcare professionals will be asked about their practices of delivering smoking cessation advice at the end of the training workshops
Practices of delivering smoking cessation advice in trained healthcare professionals at the 3-month follow-up | at the 3-month follow-up
  The trained healthcare professionals will be asked about their practices of delivering smoking cessation advice at the 3-month follow-up
Practices of delivering smoking cessation advice in trained healthcare professionals at the 6-month follow-up | at the 6-month follow-up
  The trained healthcare professionals will be asked about their practices of delivering smoking cessation advice at the 6-month follow-up
Level of self-efficacy in trained healthcare professionals before the training workshops | baseline
  The trained healthcare professionals will be asked about their levels of self-efficacy to deliver smoking cessation advice prior to the training workshops
Level of self-efficacy in trained healthcare professionals at the end of the training workshops | up to 1 week
  The trained healthcare professionals will be asked about their levels of self-efficacy to deliver smoking cessation advice at the end of the training workshops
Level of self-efficacy in trained healthcare professionals at the 3-month follow-up | at the 3-month follow-up
  The trained healthcare professionals will be asked about their levels of self-efficacy to deliver smoking cessation advice at the 3-month follow-up
Level of self-efficacy in trained healthcare professionals at the 6-month follow-up | at the 6-month follow-up
  The trained healthcare professionals will be asked about their levels of self-efficacy to deliver smoking cessation advice at the 6-month follow-up
Intention to deliver smoking cessation advice in trained healthcare professionals before the training workshops | baseline
  The trained healthcare professionals will be asked about their intentions to deliver smoking cessation advice prior to the training workshops
Intention to deliver smoking cessation advice in trained healthcare professionals at the end of the training workshops | up to 1 week
  The trained healthcare professionals will be asked about their intentions to deliver smoking cessation advice at the end of the training workshops
Intention to deliver smoking cessation advice in trained healthcare professionals aat the 3-month follow-up | at the 3-month follow-up
  The trained healthcare professionals will be asked about their intentions to deliver smoking cessation advice at the 3-month follow-up
Intention to deliver smoking cessation advice in trained healthcare professionals aat the 6-month follow-up | at the 6-month follow-up
  The trained healthcare professionals will be asked about their intentions to deliver smoking cessation advice at the 6-month follow-up
Planning to deliver smoking cessation advice in trained healthcare professionals before the training workshops | baseline
  The trained healthcare professionals will be asked about their planning to deliver smoking cessation advice prior to the training workshops
Planning to deliver smoking cessation advice in trained healthcare professionals at the end of the training workshops | up to 1 week
  The trained healthcare professionals will be asked about their planning to deliver smoking cessation advice at the end of the training workshops
Planning to deliver smoking cessation advice in trained healthcare professionals at the 3-month follow-up | at the 3-month follow-up
  The trained healthcare professionals will be asked about their planning to deliver smoking cessation advice at the 3-month follow-up
Planning to deliver smoking cessation advice in trained healthcare professionals at the 6-month follow-up | at the 6-month follow-up
  The trained healthcare professionals will be asked about their planning to deliver smoking cessation advice at the 6-month follow-up
Number of smokers that have been approached by healthcare professionals at the end of the project | at 22 months
  The numbers of smokers that have been approached by the trained healthcare professionals at the end of the project will be recorded.
Number of smokers that have been given brief advice on smoking cessation at the end of the project | at 22 months
  The numbers of smokers that have been given brief advice on smoking cessation at the end of the project will be recorded.
Number of smokers that have been referred to smoking cessation services at the end of the project | at 22 months
  The numbers of smokers that have been referred to smoking cessation services at the end of the project will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator

REFERENCES:
- [Derived] Li HCW, Xia W, Li L, Chen H, Ho LLK, Cheung KY, Xiao S, Chan YC, Chung OKJ. Evidence-based brief cessation advice plus active referral for emergency department patients who smoke: a single-arm, real-world clinical trial. BMC Med. 2025 Nov 27;23(1):714. doi: 10.1186/s12916-025-04534-9. PMID 41310683